CLINICAL TRIAL: NCT04133844
Title: Evaluation of Antithrombin Deficiency in Patients of Intensive Care Unit Placed on Extracorporeal Membrane Oxygenation
Acronym: ATECMO
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_9727_ATECMO
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Severe Cardiac Insufficiency
Keywords: extracorporeal membrane oxygenation
MeSH Terms: conditions — Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extracorporeal membrane oxygenation
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample collection from a peripheral catheter at ECMO initiation (H0), then 2h, 6h, 12h, 24h and daily from day 2 to day 7 or at ECMO discontinuation

SUMMARY:
Prospective, monocentric, non-interventional study in patients placed on extracorporeal membrane oxygenation (ECMO)

DETAILED DESCRIPTION:
Our hypothesis is that ECMO initiation is responsible for a severe decrease of antithrombin level in a high proportion of patients who develop heparin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Any ICU patient of receiving veno-arterial extracorporeal membrane oxygenation
* Patients who have not expressed opposition to participate

Exclusion Criteria:

* Arterial thrombosis or progressive venous thrombosis
* Contraindication to heparin
* Constitutional deficiency in antithrombin
* Patient refusal
* Minor patient
* Protected major (safeguard justice, trusteeship and guardianship) and persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cardiac insifficiency placed on extracorporeal membrane oxygenation (ECMO)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
To study antithrombin level from during the first 24h after ECMO initiation | Day 7
  Blood sample at ECMO initiation (H0), then 2h, 6h, 12h, 24h and daily from day 2 to day 7 or at ECMO discontinuation

SECONDARY OUTCOMES:
To study antithrombin level 24h after initialization of ECMO | Hour 24
  Blood sample at 24h
To study the prevalence of antithrombin (AT) deficiency (≤70%) at each time point (from H0 to day 7) | Day 7
  Blood sample
To study relationship between antithrombin level and heparin resistance | Day 7
  Blood sample
To study relationship between antithrombin level and thrombin generation test | Day 7
  Blood sample
To study clinical factors associated with AT deficiency | Day 7
  Blood sample
To describe clinical evolution of patients according to initial AT level | Hour 0
  Blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France